CLINICAL TRIAL: NCT02435433
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of Ramucirumab and Best Supportive Care (BSC) Versus Placebo and BSC as Second-Line Treatment in Patients With Hepatocellular Carcinoma and Elevated Baseline Alpha-Fetoprotein (AFP) Following First-Line Therapy With Sorafenib
Brief Title: A Study of Ramucirumab (LY3009806) Versus Placebo in Participants With Hepatocellular Carcinoma and Elevated Baseline Alpha-Fetoprotein
Acronym: REACH-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15755; I4T-MC-JVDE (Other: Eli Lilly and Company); 2014-005068-13 (EudraCT Number)
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ramucirumab + Best Supportive Care (BSC) (Experimental): 8 milligrams per kilogram (mg/kg) ramucirumab administered as an intravenous (IV) injection on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab
- Placebo + BSC (Placebo Comparator): Placebo administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: Placebo
- Open Label Ramucirumab + BSC (Experimental): 8 mg/kg ramucirumab administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab
- Ramucirumab MEE Cohort + BSC (Experimental): 8 mg/kg ramucirumab administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab
- Placebo MEE Cohort + BSC (Placebo Comparator): Placebo administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: Placebo

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: Cyramza; LY3009806
Drug: Placebo — Administered IV
  Arms: Placebo + BSC; Placebo MEE Cohort + BSC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ramucirumab in participants with hepatocellular carcinoma (HCC) and elevated baseline alpha-fetoprotein. Participants will be randomized to ramucirumab or placebo in a 2:1 ratio (Main Global Cohort and China Maximized Extended Enrollment [MEE] Cohort). Participants may also receive ramucirumab if eligible to be enrolled in Open-Label Expansion (OLE) Cohort.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of HCC based on histopathologic findings, or a diagnosis of cirrhosis and a tumor with classical HCC imaging characteristics.
* Sorafenib was the only systemic therapy for HCC and was discontinued for disease progression or intolerance (Main Global and MEE Cohorts only).
* The participant received ≤2 prior systemic therapy regimen, excluding prior sorafenib or chemotherapy, for the treatment of HCC (OLE Cohort only).
* ≥1 measurable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 that has not been previously treated with locoregional therapy. A participant with a lesion(s) that has previously been treated with locoregional therapy is also eligible, if the lesion has documented progression after locoregional treatment and is measureable.
* Child-Pugh score <7 (Child-Pugh Class A).
* Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy.
* Baseline AFP ≥400 nanograms/milliliter.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Resolution of all clinically significant toxic effects of prior therapy.
* Total bilirubin ≤1.5 times upper limit of normal value (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤5 × ULN.
* Creatinine clearance ≥60 milliliters/minute.
* Urinary protein is ≤1+ on dipstick or routine urinalysis or 24-hour urine demonstrating <1 gram of protein.
* Absolute neutrophil count ≥1.0 × 10^9/Liter, hemoglobin ≥9 grams/deciliter, and platelets ≥75 × 10^9/Liter.
* International Normalized Ratio (INR) ≤1.5 and a partial thromboplastin time (PTT) ≤5 seconds above the ULN.
* Surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method.
* If a woman of childbearing potential, a negative serum pregnancy test prior to randomization.
* Willing to provide blood for research. The participant has provided signed informed consent prior to any study specific procedures and is amenable to compliance with protocol schedules and testing.

Exclusion Criteria:

* Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma.
* Concurrent malignancy. Participants with carcinoma in situ of any origin and participants with prior malignancies in remission may be eligible with sponsor approval.
* Previous brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression.
* History of or current hepatic encephalopathy or clinically meaningful ascites.
* Ongoing or recent hepatorenal syndrome.
* Liver transplant (Main Global and MEE cohorts only; Participants with prior liver transplant may be eligible for OLE cohort).
* Hepatic locoregional therapy following prior systemic therapy or within 28 days prior to randomization.
* Major surgical procedure, traumatic injury, non-healing wound, or peptic ulcer ≤28 days prior to randomization.
* Received radiation to any nonhepatic (for example, bone) site within 14 days prior to randomization.
* Placement of a subcutaneous venous access device within 7 days prior to the first dose of study treatment unless the procedure is judged of low risk of bleeding.
* Enrolled in a clinical trial involving an investigational product or unapproved use of a drug or in medical research judged not to be scientifically or medically compatible with this study.
* Discontinued from study treatment from another clinical trial within 28 days prior to randomization.
* Known allergy to any of the treatment components.
* Uncontrolled hypertension.
* Any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, <6 months prior to randomization.
* Any bleeding episode considered life-threatening, or any Grade 3 or 4 gastrointestinal bleeding episode in the 3 months prior to randomization requiring intervention.
* Esophageal or gastric varices that require intervention or represent high bleeding risk. Participants with evidence of portal hypertension or prior bleeding must have had endoscopic evaluation within 3 months prior to randomization.
* Gastrointestinal perforation or fistulae within 6 months prior to randomization.
* Symptomatic congestive heart failure (New York Heart Association II-IV), unstable angina pectoris, or symptomatic or poorly controlled cardiac arrhythmia.
* Pregnant or breast-feeding.
* Any medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results. Conditions include but are not limited to:

  * Human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness.
  * Active or uncontrolled clinically serious infection. (Participants with chronic viral hepatitis are eligible.)
  * Ongoing or recent history of drug abuse.
  * Uncontrolled hereditary or acquired thrombotic or bleeding disorder.
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection.
* Therapeutic dose anticoagulation with warfarin, low molecular-weight heparin, or similar agents.
* Chronic therapy with nonsteroidal anti-inflammatory agents or other anti-platelet agents. Aspirin at doses up to 100 milligrams/day is permitted.
* The participant received prior immunotherapy and is experiencing or has experienced any of the following (OLE cohort only):

  * Any clinically significant Grade ≥3 immune-related adverse event (irAE)
  * Any grade neurologic or ocular irAE
  * Any grade immune-related pneumonitis, cardiomyopathy, or hepatitis
* The participant received prior immunotherapy and at the time of study enrollment, requires steroids or other immunosuppressive agents (OLE cohort only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours EST), Study Director — Eli Lilly and Company
Locations (120):
- United States (8):
  - Pacific Hematology and Oncology Associates, Daly City, California
  - UCLA Medical Center, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Iowa Hospital, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - OREGON HEALTH and SCIENCE UNIVERSITY, Portland, Oregon
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kurralta Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodville
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Brazil (6):
  - Fundação PIO XII, Barretos
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Barretos
  - Cenantron - Centro Avançado de Tratamento Oncológico, Belo Horizonte
  - Associação Hospital de Caridade Ijuí, Ijuí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- China (22):
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Changsha
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangdong
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Guangzhou
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Hangzhou
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Hebei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heilongjiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Henan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hubei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Nanning
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Qingdao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Shanghai
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Xi'an
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- France (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avignon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clermont-Ferrand
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
- Germany (11):
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Bayern
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Hong Kong (5):
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Hong Kong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hong Kong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kowloon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shatin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuenmen
- Israel (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benevento
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cremona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (15):
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Fukuoka
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Iizuka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanazawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kashiwa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Matsuyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shimotsuke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suita-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunto-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yokohama
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
- Spain (4):
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bern, Switzerland
- Taiwan (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buzi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Acton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bebington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Shao G, Bai Y, Yuan X, Chen X, Gu S, Gu K, Hu C, Liang H, Guo Y, Wang J, Yen CJ, Lee VH, Wang C, Widau RC, Zhang W, Liu J, Zhang Q, Qin S. Ramucirumab as second-line treatment in Chinese patients with advanced hepatocellular carcinoma and elevated alpha-fetoprotein after sorafenib (REACH-2 China): A randomised, multicentre, double-blind study. EClinicalMedicine. 2022 Oct 6;54:101679. doi: 10.1016/j.eclinm.2022.101679. eCollection 2022 Dec. PMID 36247923
- [Derived] Llovet JM, Singal AG, Villanueva A, Finn RS, Kudo M, Galle PR, Ikeda M, Callies S, McGrath LM, Wang C, Abada P, Widau RC, Gonzalez-Gugel E, Zhu AX. Prognostic and Predictive Factors in Patients with Advanced HCC and Elevated Alpha-Fetoprotein Treated with Ramucirumab in Two Randomized Phase III Trials. Clin Cancer Res. 2022 Jun 1;28(11):2297-2305. doi: 10.1158/1078-0432.CCR-21-4000. PMID 35247922
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Trojan J, Mollon P, Daniele B, Marteau F, Martin L, Li Y, Xu Q, Piscaglia F, Zaucha R, Sarker D, Lim HY, Venerito M. Comparative Efficacy of Cabozantinib and Ramucirumab After Sorafenib for Patients with Hepatocellular Carcinoma and Alpha-fetoprotein >/= 400 ng/mL: A Matching-Adjusted Indirect Comparison. Adv Ther. 2021 May;38(5):2472-2490. doi: 10.1007/s12325-021-01700-2. Epub 2021 Apr 6. PMID 33822328
- [Derived] Zhu AX, Finn RS, Kang YK, Yen CJ, Galle PR, Llovet JM, Assenat E, Brandi G, Motomura K, Ohno I, Daniele B, Vogel A, Yamashita T, Hsu CH, Gerken G, Bilbruck J, Hsu Y, Liang K, Widau RC, Wang C, Abada P, Kudo M. Serum alpha-fetoprotein and clinical outcomes in patients with advanced hepatocellular carcinoma treated with ramucirumab. Br J Cancer. 2021 Apr;124(8):1388-1397. doi: 10.1038/s41416-021-01260-w. Epub 2021 Feb 3. PMID 33531690
- [Derived] Reig M, Galle PR, Kudo M, Finn R, Llovet JM, Metti AL, Schelman WR, Liang K, Wang C, Widau RC, Abada P, Zhu AX. Pattern of progression in advanced hepatocellular carcinoma treated with ramucirumab. Liver Int. 2021 Mar;41(3):598-607. doi: 10.1111/liv.14731. Epub 2020 Dec 5. PMID 33188713
- [Derived] Zhu AX, Nipp RD, Finn RS, Galle PR, Llovet JM, Blanc JF, Okusaka T, Chau I, Cella D, Girvan A, Gable J, Bowman L, Wang C, Hsu Y, Abada PB, Kudo M. Ramucirumab in the second-line for patients with hepatocellular carcinoma and elevated alpha-fetoprotein: patient-reported outcomes across two randomised clinical trials. ESMO Open. 2020 Aug;5(4):e000797. doi: 10.1136/esmoopen-2020-000797. PMID 32817068
- [Derived] Kudo M, Okusaka T, Motomura K, Ohno I, Morimoto M, Seo S, Wada Y, Sato S, Yamashita T, Furukawa M, Aramaki T, Nadano S, Ohkawa K, Fujii H, Kudo T, Furuse J, Takai H, Homma G, Yoshikawa R, Zhu AX. Ramucirumab after prior sorafenib in patients with advanced hepatocellular carcinoma and elevated alpha-fetoprotein: Japanese subgroup analysis of the REACH-2 trial. J Gastroenterol. 2020 Jun;55(6):627-639. doi: 10.1007/s00535-020-01668-w. Epub 2020 Feb 27. PMID 32107609
- [Derived] Zhu AX, Kang YK, Yen CJ, Finn RS, Galle PR, Llovet JM, Assenat E, Brandi G, Pracht M, Lim HY, Rau KM, Motomura K, Ohno I, Merle P, Daniele B, Shin DB, Gerken G, Borg C, Hiriart JB, Okusaka T, Morimoto M, Hsu Y, Abada PB, Kudo M; REACH-2 study investigators. Ramucirumab after sorafenib in patients with advanced hepatocellular carcinoma and increased alpha-fetoprotein concentrations (REACH-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Feb;20(2):282-296. doi: 10.1016/S1470-2045(18)30937-9. Epub 2019 Jan 18. PMID 30665869
- See also: A Study of Ramucirumab (LY3009806) Versus Placebo in Participants With Hepatocellular Carcinoma and Elevated Baseline Alpha-Fetoprotein — https://trials.lillytrialguide.com/en-US/trial/12euK0N4aQe2aiGqC6GEQ4

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Main study: Participants who received sorafenib as first-line therapy were randomized to ramucirumab or placebo.
  2. Open-Label Expansion: Participants who were not previously treated with sorafenib were enrolled into this single-arm addenda and treated with ramucirumab. The purpose of this addenda is to monitor safety, and data was reported under AE section.
  (Continued...)
Pre-assignment Details: c. China Maximized Extended Enrollment: This is an extension phase of the main study, with an additional 60 participants enrolled in China. Safety was monitored and data was reported under AE section.
Groups:
- Ramucirumab + BSC: 8 milligrams per kilogram (mg/kg) ramucirumab administered as an intravenous (IV) injection on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
- Ramucirumab MEE Cohort: 8 mg/kg ramucirumab administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
- Placebo MEE Cohort: Placebo administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Ramucirumab + BSC | Placebo + BSC | Open Label Ramucirumab + BSC | Ramucirumab MEE Cohort | Placebo MEE Cohort
Started | 197 | 95 | 47 | 39 | 21
Participants Who Received Study Drug | 197 | 95 | 47 | 39 | 21
Completed (Completers include participants who had died due to any cause or alive and on study at the end of study, but off treatment.) | 193 | 90 | 42 | 38 | 21
Not Completed | 4 | 5 | 5 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Ramucirumab + BSC: 8 mg/kg ramucirumab administered as an IV injection on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
- Placebo + Best Supportive Care (BSC); Placebo MEE Cohort: Placebo administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Participants still on treatment at the time of study completion may have the option to crossover to the ramucirumab arm.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + BSC | Placebo + Best Supportive Care (BSC) | Open Label Ramucirumab + BSC | Ramucirumab MEE Cohort | Placebo MEE Cohort | Total
Number analyzed (Participants) | 197 | 95 | 47 | 39 | 21 | 399
Age, Continuous [Median (Full Range); unit: years] | 64 [30 to 88] | 64 [26 to 85] | 61 [36 to 82] | 54 [24 to 74] | 54 [31 to 66] | 62 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 16 | 6 | 7 | 1 | 73
  Male | 154 | 79 | 41 | 32 | 20 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 1 | 0 | 0 | 22
  Not Hispanic or Latino | 129 | 58 | 40 | 12 | 9 | 248
  Unknown or Not Reported | 56 | 28 | 6 | 27 | 12 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 102 | 45 | 26 | 39 | 21 | 233
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 4 | 0 | 0 | 6
  White | 60 | 31 | 13 | 0 | 0 | 104
  More than one race | 0 | 1 | 4 | 0 | 0 | 5
  Unknown or Not Reported | 34 | 17 | 0 | 0 | 0 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 6 | 1 | 8 | 0 | 0 | 15
  United States | 10 | 1 | 12 | 0 | 0 | 23
  Czechia | 4 | 2 | 0 | 0 | 0 | 6
  Japan | 41 | 18 | 0 | 0 | 0 | 59
  United Kingdom | 9 | 2 | 0 | 0 | 0 | 11
  Switzerland | 2 | 2 | 1 | 0 | 0 | 5
  Spain | 3 | 2 | 0 | 0 | 0 | 5
  Canada | 1 | 1 | 0 | 0 | 0 | 2
  Austria | 1 | 1 | 0 | 0 | 0 | 2
  South Korea | 24 | 14 | 0 | 0 | 0 | 38
  Belgium | 2 | 2 | 0 | 0 | 0 | 4
  China | 3 | 1 | 8 | 39 | 21 | 72
  Taiwan | 22 | 11 | 10 | 0 | 0 | 43
  Brazil | 5 | 4 | 0 | 0 | 0 | 9
  Poland | 2 | 3 | 0 | 0 | 0 | 5
  Italy | 13 | 9 | 0 | 0 | 0 | 22
  Israel | 1 | 0 | 0 | 0 | 0 | 1
  Australia | 2 | 1 | 0 | 0 | 0 | 3
  France | 34 | 17 | 0 | 0 | 0 | 51
  Germany | 12 | 3 | 8 | 0 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS time was measured from date of randomization to date of death from any cause. Participants who were not known to have died on or before the date of data cut-off, OS data was censored on the last date (on or before the cut-off date) the participant was known to be alive.
Time Frame: From Date of Randomization to Death from Any Cause (Up to 28 Months)
Population: All randomized participants. Participants were censored in Ramucirumab arm = 50 and Placebo arm = 21. All randomized participants (including the censored participants) were included in the analyses.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo + BSC: Placebo administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Participants still on treatment at the time of study completion may have the option to crossover to the ramucirumab arm.
Arm/Group | Ramucirumab + Best Supportive Care (BSC) | Placebo + BSC
Number analyzed (Participants) | 197 | 95
Months | 8.51 [7.00 to 10.58] | 7.29 [5.42 to 9.07]
Statistical Analysis 1: Comparison: Ramucirumab + Best Supportive Care (BSC) vs Placebo + BSC; Test type: Superiority; p = 0.0199, Log Rank; Hazard Ratio (HR) = 0.710, 95% CI 2-sided [0.531 to 0.949] — Stratified analysis

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival is defined as time from the date of randomization to the date of first observation of objective progression or death from any cause.
Time Frame: From Randomization to Objective Progression or Death from Any Cause (Up to 28 Months)
Population: All randomized participants. Participants were censored in the Ramucirumab arm = 25 and in the Placebo arm = 9. All randomized participants (including the censored participants) were included in the analyses.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ramucirumab + BSC: 8 mg/kg ramucirumab administered as an intravenous IV injection on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 197 | 95
Months | 2.83 [2.76 to 4.11] | 1.61 [1.45 to 2.69]
Statistical Analysis 1: Comparison: Ramucirumab + BSC vs Placebo + BSC; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.452, 95% CI 2-sided [0.339 to 0.603] — Stratified analysis

3. Secondary Outcome: Time to Radiographic Progression
Description: Time to radiographic progression is defined as the time from the date of randomization to the date of first observation of objective progression.
Time Frame: From Randomization to Objective Progression (Up to 28 Months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 197 | 95
Months | 3.02 [2.79 to 4.17] | 1.61 [1.45 to 2.73]
Statistical Analysis 1: Comparison: Ramucirumab + BSC vs Placebo + BSC; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.427, 95% CI 2-sided [0.313 to 0.582] — Stratified analysis

4. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR): Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants who achieve a best overall response of complete response (CR) + partial response (PR). ORR = CR + PR. CR is the disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. Best overall response is classified based on the overall responses assessed by study investigators according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Time Frame: From Randomization to Objective Progression (Up to 28 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 197 | 95
percentage of participants | 4.6 | 1.1
Statistical Analysis 1: Comparison: Ramucirumab + BSC vs Placebo + BSC; Test type: Superiority; p = 0.1697, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.6, 95% CI 2-sided [0.6 to 37.3] — Stratified analysis

5. Secondary Outcome: Pharmacokinetics (PK): Minimum Serum Concentration (Cmin) Before 2nd, 4th, 7th, and 10th Infusion
Description: PK Cmin of Ramucirumab Blood samples were collected at specified time points, and in the event of an infusion-related reaction, for assessment of ramucirumab serum concentrations.
Time Frame: Predose, Weeks 2, 6, 12 and 18, Day 1; Up to 3 Days Before Infusion (14-Day Cycles)
Population: All randomized participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Ramucirumab + BSC
Number analyzed (Participants) | 195
nanogram/milliliter (ng/mL)
  Week 0 | NA (NA) — 1 trough concentrations that was reported below the limit of quantitation were treated as missing for the concentration summaries.
  Week 2 | 23.5 (57)
  Week 6 | 44.1 (60)
  Week 12 | 60.2 (46)
  Week 18 | 63.2 (40)

6. Secondary Outcome: PK: Serum Concentration Maximum (Cmax) After 1st, 2nd, 4th, 7th and 10th Ram Infusion
Description: PK Cmax of Ramucirumab Blood samples were collected at specified time points, and in the event of an infusion-related reaction, for assessment of ramucirumab serum concentrations.
Time Frame: Weeks 0, 2, 6, 12 and 18, Day 1; 1 hour to 1.5 hours Post End of Infusion (14 day-Cycles)
Population: All randomized participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ramucirumab + BSC
Number analyzed (Participants) | 195
ng/mL
  Week 0 | 156 (22)
  Week 2 | 181 (24)
  Week 6 | 205 (24)
  Week 12 | 221 (24)
  Week 18 | 228 (22)

7. Secondary Outcome: Percentage of Participants With Anti-Ramucirumab Antibodies
Description: Percentage of participants with positive treatment emergent anti-drug antibodies was summarized by treatment group. A treatment-emergent ADA (TEADA) was defined as: having a negative ADA at baseline and an ADA titer greater than or equal to 1:20 (that is (i.e.), greater than 2-fold from the minimal required dilution of 1:10) any time post baseline (i.e., treatment-induced); or a 4-fold or greater change in ADA titer from baseline for participants that had a detectable ADA titer at baseline (i.e., treatment boosted).
Time Frame: Predose Cycle 1: 7 Days prior to First Infusion, Cycle 4: 3 Days Prior to Infusion, Cycle 7 through Follow Up (Up to 28 Months)
Population: All randomized participants who received at least one dose of study drug and had evaluable anti-ramucirumab data.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 161 | 76
percentage of participants | 5.0 | 9.2

8. Secondary Outcome: Time to Deterioration of Functional Assessment of Cancer Therapy (FACT) Hepatobiliary Symptom Index-8 (FHSI-8)
Description: The FACT Hepatobiliary Symptom Index (FHSI-8) is a instrument with specific focus regarding the most frequent and concerning symptoms experienced by participants with hepatobiliary malignancies, including lack of energy, nausea, pain, weight loss, pain in back, fatigue, jaundice, stomach pain or discomfort. The (FHSI-8) questionnaire was used to assess the time to deterioration of FSHI-8 total score issued from the date of randomization to the first date observing deterioration, with the deterioration threshold defined as a decrease ≥ 3-points from baseline. In case of no deterioration, the participants were censored at the time of the last FSHI-8 item recording. FHSI-8 total score ranges from 0 to 32 where "0" is a severely symptomatic participant and the highest score indicates an asymptomatic participant. Kaplan-Meier method Hazard ratio was used to estimate (Ramucirumab versus Placebo) and 95% Confidence Interval (CI) (Wald) were estimated from un-stratified/stratified Cox model.
Time Frame: From Randomization to the First Date of Deterioration Observation (≥ 3-point decrease) (Up to 28 Months)
Population: All randomized participants who had evaluable FHSI-8 data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 197 | 95
Months | 3.71 [2.79 to 4.40] | 2.79 [1.64 to 2.89]
Statistical Analysis 1: Comparison: Ramucirumab + BSC vs Placebo + BSC; Test type: Superiority; p = 0.2382, Log Rank; Hazard Ratio (HR) = 0.799, 95% CI 2-sided [0.545 to 1.171] — Stratified analysis

9. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire
Description: The EQ-5D-5L is a nonspecific and standardized instrument for use as a measure of self-reported health status (EuroQol Group 1990; Herdman et al. 2011). Participants completed the 5-level (no problems, slight problems, moderate problems, severe problems, and extreme problems), 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) questionnaire concerning their current health state. A unique EQ-5D-5L health state scale ranges from 0 to 100 and is defined by combining 1 level from each of the 5 dimensions. Participants indicated their current health status by marking on a continuum ranging from 100 (best imaginable health state) to 0 (worst imaginable health state).
Time Frame: From Randomization through End of Study (Up to 28 Months)
Population: All randomized participants and had evaluable EQ-5D-5L data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 197 | 95
units on a scale | -0.105 (0.201) | -0.099 (0.170)

10. Secondary Outcome: Time to Deterioration in Eastern Cooperative Oncology Group Performance Status (ECOG PS)
Description: Time to deterioration in ECOG PS is defined as the time from the date of randomization to the first date observing ECOG PS 2 (ie, deterioration from baseline status of 0 [fully active] or 1 [restricted in physically strenuous activity but ambulatory and able to carry out light work]). Participants without PS deterioration were censored at their last documented assessments of 0 or 1. Assessments included ECOG Performance Status (PS): 2- Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours, 3 -Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours, 4 -Completely disabled, cannot carry on any self-care. Totally confined to bed or chair, 5- Dead.
Time Frame: From Randomization through First Date of Deterioration Observation (ECOG PS≥2) (Up to 28 Months)
Population: All randomized participants and had evaluable ECOG data. Censored participants without any post baseline assessments at randomization date were in the Ramucirumab + BSC arm = 141 and the Placebo + BSC arm =75. All randomized participants (including the censored participants) were included in the analyses.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + BSC | Placebo + BSC
Number analyzed (Participants) | 197 | 95
Months | NA [9.33 to NA] — The median and upper limit 95% confidence interval upper limit had insufficient events to perform a meaningful statistical evaluation. | NA [5.26 to NA] — The median and upper limit 95% confidence interval had insufficient events to perform a meaningful statistical evaluation.

ADVERSE EVENTS:
Time Frame: Baseline up to 3.2 years
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo+BSC; Placebo MEE Cohort: Placebo administered IV on day 1 of each 14 day cycle. Participants may continue treatment until discontinuation criteria are met.
  Participants still on treatment at the time of study completion may have the option to crossover to the ramucirumab arm.
Arm/Group | Ramucirumab + BSC | Placebo+BSC | Open Label Ramucirumab + BSC | Ramucirumab MEE Cohort | Placebo MEE Cohort
All-Cause Mortality (participants affected / at risk) | 162/197 | 76/95 | 33/47 | 35/39 | 18/21
Serious Adverse Events (participants affected / at risk) | 72/197 | 27/95 | 18/47 | 10/39 | 3/21
Other Adverse Events (participants affected / at risk) | 189/197 | 77/95 | 40/47 | 39/39 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + BSC (N=197) | Placebo+BSC (N=95) | Open Label Ramucirumab + BSC (N=47) | Ramucirumab MEE Cohort (N=39) | Placebo MEE Cohort (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 3 (4) | 2 (3) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration pleural cavity (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma hepatic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis migrans (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + BSC (N=197) | Placebo+BSC (N=95) | Open Label Ramucirumab + BSC (N=47) | Ramucirumab MEE Cohort (N=39) | Placebo MEE Cohort (N=21)
Anaemia (Blood and lymphatic system disorders) | 19 (28) | 6 (7) | 4 (5) | 7 (13) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (16) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 16 (18) | 5 (6) | 4 (4) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 36 (46) | 12 (16) | 4 (4) | 7 (10) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 34 (47) | 7 (7) | 6 (6) | 7 (8) | 2 (2)
Constipation (Gastrointestinal disorders) | 27 (33) | 18 (19) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 33 (46) | 14 (18) | 9 (13) | 2 (3) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 37 (47) | 10 (12) | 6 (6) | 4 (4) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 20 (24) | 7 (7) | 4 (5) | 3 (4) | 3 (3)
Asthenia (General disorders) | 17 (41) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 5 (6) | 1 (2) | 1 (1) | 0 (0)
Face oedema (General disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Fatigue (General disorders) | 54 (79) | 16 (23) | 7 (8) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 10 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 16 (19) | 5 (6) | 0 (0) | 5 (12) | 0 (0)
Oedema (General disorders) | 6 (6) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 52 (69) | 13 (13) | 7 (10) | 6 (13) | 2 (2)
Pyrexia (General disorders) | 19 (23) | 3 (3) | 3 (3) | 6 (8) | 3 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (5) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (18) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (12) | 5 (6) | 2 (3) | 8 (12) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 16 (27) | 10 (15) | 3 (3) | 15 (22) | 7 (9)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (2) | 3 (4) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 21 (39) | 8 (16) | 5 (5) | 11 (27) | 6 (12)
Blood creatinine increased (Investigations) | 9 (15) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 5 (6) | 2 (3) | 3 (3) | 5 (6)
Neutrophil count decreased (Investigations) | 12 (30) | 0 (0) | 1 (2) | 6 (8) | 3 (6)
Platelet count decreased (Investigations) | 23 (72) | 2 (3) | 6 (22) | 14 (27) | 0 (0)
Urinary occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 1 (1)
Weight decreased (Investigations) | 22 (25) | 6 (7) | 2 (6) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 7 (26) | 0 (0) | 2 (3) | 6 (10) | 2 (3)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 49 (60) | 19 (19) | 6 (6) | 3 (3) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (21) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (29) | 4 (4) | 4 (7) | 14 (24) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (16) | 1 (1) | 4 (7) | 3 (9) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (21) | 5 (7) | 3 (3) | 2 (3) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (23) | 7 (8) | 2 (2) | 2 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 9 (10) | 8 (8) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 28 (36) | 5 (5) | 1 (1) | 2 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 21 (24) | 6 (8) | 3 (3) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 43 (74) | 4 (4) | 12 (21) | 10 (16) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 6 (7) | 5 (6) | 4 (4) | 4 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 8 (9) | 3 (3) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (16) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 14 (19) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 50 (79) | 12 (13) | 11 (16) | 7 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT02435433/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02435433/SAP_001.pdf